CLINICAL TRIAL: NCT04323345
Title: The Efficacy of Natural Honey in Patients Infected With Novel Coronavirus (COVID-19) : A Randomized, Controlled ,Single Masked , Investigator Initiated, Multi-center Trial
Brief Title: Efficacy of Natural Honey Treatment in Patients With Novel Coronavirus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Tantawy, Consultant Cardiologist, Sr. Researcher, Health Strategist, Health Economist & Administrator, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUST23032020
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: Coronavirus; Natural Honey
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural Honey Group (Experimental): Natural Honey
  1gm/kg/day divided into 2 to 3 doses for 14 days in addition to standard care
  Interventions: Dietary Supplement: Natural Honey; Other: Standard Care
- Standard Care (Active Comparator): Current standard care including supportive measures and lopinavir/ritonavir tablets or Arbidol or chloroquine phosphate or Hydroxychloroquine or oseltamivir with or without azithromycin.
  Interventions: Other: Standard Care

INTERVENTIONS:
Dietary Supplement: Natural Honey — Natural Honey supplement 1gm/kg/day divided into 2 to 3 doses for 14 days either orally or through nasogastric tube.
  Arms: Natural Honey Group
Other: Standard Care — Supportive measures and lopinavir/ritonavir tablets or Arbidol or chloroquine phosphate or Hydroxychloroquine or oseltamivir with or without azithromycin.

SUMMARY:
The novel coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS CoV-2) has been discovered recently in December 2019 from wuhan city in China to spread in more than 40 countries allover the world. This disease has gain the attention of all nations after it has been stated as a pandemic by the World Health Organization (WHO) in March 12, 2020. Currently no treatment has been proved to be efficient in the treatment of infected patients by COVID-19. Natural honey has been demonstrated as potent antimicrobial in many research investigations and has been considered a good alternative for antiviral drugs for the treatment of some viral infections. The investigators aim to study the efficacy of natural honey in the treatment of COVID-19 patients in this randomized , multicenter, controlled trial, comparing honey in one arm to standard care in the other arm.

DETAILED DESCRIPTION:
The (SARS CoV-2) virus is spreading globally, threatening all healthcare systems. Many healthcare systems and organizations are using different protocols and measures to fight the COVID-19. Hydroxychloroquine, lopinavir and other antiviral medications are currently under research investigations. Natural honey has been well known for its high health properties in diabetes, nutrition, dyslipidemia, skin lesions and it got FDA approval for topical wound treatment in 2007 as the most potent antimicrobial agent. Honey has been previously considered as an alternative for acyclovir in the treatment of herpes simplex virus 1 (HSV-1) and it also demonstrated for its significant antiviral effect against varicella zoster virus (VZV). Many studies have demonstrated the broad spectrum antimicrobial effect of honey as an antibacterial, anti fungal, antiviral and antimycobacterial. The National Institute for Health and Care Excellence (NICE) and the Public Health England (PHE) guidelines recommended honey as a first line of treatment for acute cough caused by upper respiratory tract infection which is currently a cornerstone symptom in COVID-19 infectious disease. Moreover, natural honey should no longer be used as "alternative" and deserves to gain more attention by scientists and researchers. The aim of this trial is to study the efficacy of natural honey in treatment of patients infected with COVID-19 in comparison with current standard care.

Methods:

This will be a randomized , multi center, double armed clinical trial, patients will be randomly assigned to two groups on 1:1 basis. Natural honey group will include patients receiving standard care and added intervention in the form of natural honey in a dose of 1gm/kg/day (previously used safely in small studies) divided into 2 to 3 doses for continuous 14 days. The other arm is the arm receiving the standard care according to the center protocol.

Our primary outcome is days for recovery using the parameters: turning from positive to negative swaps, days from fever to no fever and lung inflammation recovery in x ray or CT, our secondary outcome is the 30 days mortality rate. Data will be collected and statistically managed using STATA blindly from who received the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the criteria for diagnosis of COVID-19, either clinically or as confirmed by positive swap.

Exclusion Criteria:

* Children below 5 years old. Severely ill patients with either terminal disease. Nil per os (NPO) patients with contraindication to nasogastric tube feeding.

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Rate of recovery from positive to negative swaps | 14 days
  Percentage of patients turned from positive to negative swaps at day 14
Fever to normal temperature in days | 14 days
  Number of days till no fever
Resolution of lung inflammation in CT or X ray | 30 days
  Number of days till lungs recovery in chest X ray or CT

SECONDARY OUTCOMES:
30 days mortality rate | 30 days
  mortality rate in each group at 30 days
Number of days till reaching negative swab results | 30 days
  Number of days from initiation of intervention till changing of the swap test result from positive to negative

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Tantawy, MD, Study Chair — Misr University for Science and Technology
Locations (1):
- Mahmoud Tantawy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Honey for acute cough in children — https://www.ncbi.nlm.nih.gov/pubmed/22419319
- See also: NICE Guidelines (NG120) — https://www.nice.org.uk/guidance/ng120/chapter/Summary-of-the-evidence
- See also: The scolicidal effects of honey — https://link.springer.com/article/10.1007%2FBF02850228
- See also: Antimicrobial properties of honey — https://doi.org/10.1097/MJT.0b013e318293b09b
- See also: In vitro antiviral activity of honey against varicella zoster virus (VZV): A translational medicine study for potential remedy for shingles — https://www.transbiomedicine.com/translational-biomedicine/in-vitro-antiviral-activity-of-honey-against-varicella-zoster-virus-vzv-a-translational-medicine-study-for-potential-remedy-for-shingles.php?aid=2493
- See also: Antiviral Activities of Honey, Royal Jelly, and Acyclovir Against HSV-1 — https://www.woundsresearch.com/article/antiviral-activities-honey-royal-jelly-and-acyclovir-against-hsv-1
- See also: Therapeutic Manuka Honey: No Longer So Alternative — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4837971/
- See also: Honey-based dressings and wound care: an option for care in the United States — https://www.ncbi.nlm.nih.gov/pubmed/?term=pieper+b+honey+based